CLINICAL TRIAL: NCT00912483
Title: Efficacy of Sodium Heparin 5.000 UI/0.25 mL (Blausiegel) Compared With Heparin Sodium 5.000 USP (APP Pharmaceuticals)for Venous Thromboembolism Prophylaxis In Surgical Patients With Medium Risk For The Thromboembolism Development
Brief Title: Efficacy of Sodium Heparin in Prophylaxis of Venous Thromboembolism in Surgical Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clinica Pesquisa e Desenvolvimento Ltda
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HEPBLA0409; Thomboembolism; Heparin; Prophylaxis
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Venous Thromboembolism
Keywords: VTE
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Heparin Sodium 5.000UI/0.25mL
  Interventions: Biological: heparin sodium - Blausiegel
- Ative comparator (Active Comparator): Heparin Sodium 5.000USP/mL
  Interventions: Biological: Heparin sodium - APP

INTERVENTIONS:
Biological: heparin sodium - Blausiegel — Heparin sodium - 5.000UI/0.25mL, twice a day for 7 days and 2 hours before the surgery
  Arms: Test
Biological: Heparin sodium - APP — Heparin sodium - 5.000USP/mL, twice a day for 7 days and 2 hours before the surgery
  Arms: Ative comparator

SUMMARY:
The Venous thromboembolism (VTE) disease is very frequent, mainly as complications of medical diseases and surgical procedures. It has high prevalence and can lead to severe complications such as pulmonary embolism and postthrombotic syndrome. Although its incidence has been decreasing in recent years, the EP and DVT is still a major public health problem, especially in advanced age.

The tracking of this disease through imaging tests in asymptomatic patients does not seem to be a cost-effective, further treatment of complications is expensive and subject to no satisfactory answers are not completely effective in regard to late complications. Therefore, according CAIAFA & BASTOS (2002), effective prophylaxis is the best strategy.

The type of prevention to be used should be based on the risk of developing VTE, ie low, medium or high. Framework for a category of risk for the indication of prophylaxis, each patient should be evaluated individually and carefully to the risk of developing VTE. Maffei et al. (2005) describe the "Standards for Clinical Guideline for the prevention, diagnosis and treatment of deep vein thrombosis." According to the guide, the concentration of heparin in 5.000UI is indicated for cases of moderate-risk surgeries. Are classified as "moderate risk" to more surgery (general, gynecological and urological) in patients 40 to 60 years without additional risk factors, and the magnitude of any surgery in patients under 40 years of age who use estrogen ( Annex 01). The dosing schedule chosen in this study also follows the recommendation of the guide and is universally used .

According to Maffei et al. (2005), the diagnosis of VTE must be initiated by the history and physical examination, and then must be performed ultrasound Doppler of lower limbs. Thus, the ultra-sonography/doppler examination will be done at the beginning and end of treatment and physical examination will be done periodically throughout the period of monitoring.

Following the guidelines proposed by the literature consulted, was established to test this methodology, which aims to demonstrate the non inferiority clinical heparin sodium 5.000UI / 0.25 mL sodium heparin on 5.000UI / 1.0 mL, both produced by Blausiegel Industry and Trade Ltda. in reducing the incidence of VTE. The two formulations are produced from the same material, but have different drug concentrations. Thus, there is a need to scientifically prove that the therapeutic activity and safety of the product test is non-inferior to the comparator drug (APP heparina - 5.000 USP/mL), allowing the sponsoring company to obtain the registration of the product in the concentration of 5000UI /0.25 mL in ANVISA at the proposed therapeutic indication in the study.

ELIGIBILITY:
Inclusion Criteria:

* Accept all items described in Informed Consent, signing it in two ways;
* Age between 40 and 60 years without additional risk factors, which held more surgery (general, gynecological and urological);
* Women aged 18 to 40 years making use of estrogen;
* Be alert to the need for surgery antithrombotic prophylaxis;
* Be classified as "moderate risk" for developing VTE, according to the protocol of prophylaxis of deep vein thrombosis of the Brazilian Society of Angiology and Vascular Surgery.

Exclusion Criteria:

* Acute coronary syndrome;
* Immobilization of the lower limbs due to fractures, because in this way will be considered as high risk;
* history of recent stroke;
* Patients at high risk of bleeding in which the use of heparin is contra-indicated;
* General Surgery in patients over 60 years in the case of patients at high risk for VTE;
* general surgery in patients 40 to 60 years with additional risk factors for development of VTE;
* Major amputations;
* more orthopedic surgeries;
* Patients with pre-surgical diagnosis of malignant neoplasms;
* Patients with a platelet level below 100x109 / L;
* Use of anticoagulants 48 hours before randomization;
* severe liver failure;
* Be classified as "Low Risk" or "high risk" for developing VTE
* Pregnancy and lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of venous thromboembolism during the 28 days of study | 2h before the start of surgery; 1 d. after 1st administration; 3 days; 5 days; 7 days; 14 days; 21 days; 28 days

SECONDARY OUTCOMES:
Incidence of adverse reactions during the treatment period | 1 d. after 1st administration; 3 days; 5 days; 7 days; 14 days; 21 days; 28 days